CLINICAL TRIAL: NCT04096937
Title: Journey of Hope in Appalachia: Supporting Resilience in the Region's Youth
Acronym: JOHA
Status: Completed | Type: Observational
Sponsor: Gia Mudd (Other)
Collaborators: West Virginia University (Other)
Responsible Party: Sponsor-Investigator, Gia Mudd, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 46776
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Adverse Childhood Experiences
Keywords: Resilience; Appalachian youth; Community-based participatory research
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Appalachian adults: Adults in Appalachia invested in well-being of youth.
  Interventions: Other: Focus groups
- Appalachian youth: Youth from 7th through 12th grade.
  Interventions: Other: Focus groups

INTERVENTIONS:
Other: Focus groups — Focus groups will be conducted with adult stakeholders and with youth in Appalachia. Feedback from the focus groups will guide cultural tailoring of the Journey of Hope in Appalachia intervention for use in a later phase.

SUMMARY:
Rural youth have heightened exposure to adverse childhood experiences (ACES) such as poverty, social isolation, chronic hunger, and drug use in the home. These threats can lead to downstream problems with emotion regulation, substance abuse, and heightened vulnerability to chronic disease. Resilience is the capacity to adapt positively in the face of such disadvantage. Youth resilience interventions can buffer the negative effects of ACES. Unfortunately, rural schools and other youth-serving agencies often have inadequate capacity to provide such interventions. Thus, there is a critical need to develop cost-effective, sustainable, and culturally-relevant youth resilience interventions that can be delivered by trained personnel with dedicated time and resources. WVU, UK, and Save The Children have a long-term goal to establish a sustained community-engaged research partnership to promote resilience in Appalachian youth. This is a community-based participatory research (CBPR)-guided study being conducted for the purpose of developing a culturally relevant, intervention to promote Appalachian youth resilience. The intervention, called Journey of Hope in Appalachia (JOHA), has as it's starting point Save The Children's evidence-based Journey of Hope (JOH) program that targets youth experiencing acute stress from natural disasters and similar events. This program will be culturally adapted to promote resilience among Appalachian youth experiencing ACES. JOHA will incorporate positive aspects of Appalachian culture (e.g., storytelling, theater, music) and will be designed for sustainability and eventual dissemination by Save through the Appalachian Translational Research Network (ATRN) and other regional Networks.

ELIGIBILITY:
Inclusion Criteria:

* Youth or adults who are residents of Appalachia
* Able to read and speak in English

Exclusion Criteria:

* Youth or adults who are not residents of Appalachia Kentucky or West Virginia
* Children under the age of 10

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Youth of Appalachia Kentucky and West Virginia and adults who are parents of youth or are stakeholders in the health and well-being of Appalachian youth.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Number of themes | 6 months
  Number of themes that emerge from the focus group data useful for guiding cultural tailoring of the Journey of Hope in Appalachia intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gia Mudd-Martin, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Center of Excellence in Rural Health, Hazard, Kentucky
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No